CLINICAL TRIAL: NCT06341439
Title: Clinical Efficacy of Mouthrinses Based on Chlorhexidine 0.12% and CITROX® as a Support to Non-surgical Periodontal Therapy: a Randomized Controlled Triple-blind Clinical Trial
Brief Title: Clinical Efficacy of Mouthrinses Based on Chlorhexidine 0.12% and CITROX®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Enrico Marchetti, Associate Professor, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Prot. 001_2023
Record Dates: First submitted 2024-03-14; First posted 2024-04-02 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis
Keywords: Periodontitis; Non-surgical therapy; Chlorhexidine; Mouthwash; Plaque; Randomized trial
MeSH Terms: conditions — Periodontitis; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Mouthwash containing 0,12% chlorhexidine + bioflavonoids
  Interventions: Device: Mouthwash with chlorhexidine 0,12% and CITROX
- Control Group (Active Comparator): Mouthwash containing 0,12% chlorhexidine
  Interventions: Device: Mouthwash with chlorhexidine 0,12%

INTERVENTIONS:
Device: Mouthwash with chlorhexidine 0,12% and CITROX — Patients use the undiluted mouthwash 2 times a day for 14 days after performing normal brushing.
  Arms: Test Group
Device: Mouthwash with chlorhexidine 0,12% — Patients use the undiluted mouthwash 2 times a day for 14 days after performing normal brushing.
  Arms: Control Group

SUMMARY:
The goal of the following clinical trial is to compare the efficacy of a product based on chlorhexidine 0.12% and CITROX and the same product without CITROX in the healing phenomena that occur after non-surgical periodontal therapy. The main questions it aims to answer are:

* Is the response to periodontal therapy better if mouthwashes containing bioflavonoids are used as a support to non surgical periodontal therapy?
* What is the patients' perception?

Participants, divided into 2 groups, are asked to use either one or the other mouthwash for 14 days after non-surgical periodontal therapy.

DETAILED DESCRIPTION:
At baseline, all participants underwent received comprehensive periodontal examination, full-mouth intraoral radiographic analysis and received oral hygiene instruction. All treatments were performed by the same experienced clinician (M.G.L.) After completing NSPT, patients were randomly assigned to the test- or control group through an online random number generator (random.org; www.random.org). Test group participants received a 300 ml bottle of mouthwash containing 0,12% CHX combined with organic acids and bioflavonoids, while the control group received a 300 ml bottle of 0.12% CHX mouthwash. Both bottles were unlabeled to prevent identification by either the patients or the clinician. All participants were instructed to rinse with the undiluted mouthwash twice daily (morning and evening) for 60 seconds over 14 days following subgingival instrumentations. This regimen aligns with the standard use of chlorhexidine mouthwashes. Oral hygiene instructions were provided after both supragingival debridement and subgingival instrumentations with additional training in the use of interdental devices as necessary.

Patients were recalled for follow-up assessments at 14 days (T2), 2 months (T3) and 6 months (T4). In these sessions, oral hygiene instructions were reinforced as needed. During the follow-up, no additional periodontal treatments were performed. Patients were subsequently enrolled in a maintenance care program, involving routine professional cleanings every 6 months. Data collected from baseline (T0) to 6 months (T4) were used for the present analysis.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and ASA II patients;
* Age > 21 years;
* Non-smokers or smokers < 5 cig/day;
* Presence of periodontal disease;
* >10 natural teeth;
* At least 2 teeth with pockets ≥5mm;
* Indications for carrying out at least one SRP (scaling and root planing) session;
* Signing of the written informed consent to participate in the study.

Exclusion Criteria:

* Severe general medical pathologies;
* Immunodeficiency states;
* Radiotherapy in the head and neck region;
* Uncontrolled diabetes or hypertension;
* Smokers >5 cigs/day;
* Impossibility to carry out homogeneous and continuous follow-up;
* Documented allergy to chlorhexidine or hyaluronic acid;
* Taking drugs that cause alterations in the gums and oral mucosa;
* Pregnancy or breastfeeding;
* Presence of removable prostheses;
* Periodontal treatment in the previous 6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Full mouth bleeding score (FMBS) | baseline, 14 days, 2 months, 6 months
  The FMBS indicate the percentage of bleeding sites out of the total.
Full mouth plaque score (FMPS) | baseline, 14 days, 2 months, 6 months
  The FMPS indicate the percentage of sites with plaque out of the total.
Probing Depth (PD) | baseline, 2 months, 6 months
  Effects on post-treatment healing: the Probing Depth was measured in mm
Gingival Index (GI) | baseline, 14 days, 2 months, 6 months
  Effects on post-treatment healing: the GI was assessed with values between 0 and 3 (0- best one, 3 worst one)
Plaque Index (PI) | baseline, 14 days, 2 months, 6 months
  Effects on post-treatment healing: the GI was assessed with values between 0 and 3 (0- best one, 3 worst one)

SECONDARY OUTCOMES:
Patient Reported Outcome Measure (PROMS) | 2 weeks post non-surgical periodontal therapy
  Visual Analogue Scale (VAS) in the form of a questionnaire to evaluate post-op pain, post-op sensitivity, taste alteration, appearance of staining and pleasantness of the mouthrinse used. The minimum value is 0 while the maximum value is 10. For all questions the best value is 0 and the worst 10, except for pleasantness.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Marchetti, DDS, MS, PhD, Principal Investigator — University of L'Aquila
Locations (1):
- University of L'Aquila, division of periodontology, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD could be available to other researchers. Data will anonymized and delivered under request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Under request.
Access Criteria: The team will have the possibility to choose if the request come from a reliable source.